CLINICAL TRIAL: NCT00593840
Title: Phase II Trial Evaluating Elimination of Radiation Therapy To Pathological N0 Neck(s) With Intensity Modulated Postoperative Radiation Therapy
Brief Title: Phase II Trial Evaluating Elimination of Radiation Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0142 / 201106342
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cancer of the Larynx
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensity modulated radiation therapy (IMRT) (Experimental): -This study provides guidelines for volume to be contoured during IMRT based on tumor site and stage of tumor site. The clinical tumor volume (CTV)1 will be treated to 66 Cy in 33 fractions or 60 Gy in 30 fractions. The CTV2 will be treated to 54 Gy in 33 fractions or 52 Gy in 30 fractions. The CTV3 will be modified based on tumor site and stage of tumor site in order to reduce volume.
  Interventions: Radiation: Intensity modulated radiation therapy

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy
  Other Names: IMRT

SUMMARY:
The purpose of this study is to determine if reducing or eliminating radiation treatment to one or both sides of the neck where there is no evidence of cancer can help spare the side effects of radiation treatment for head and neck cancer. In this study, the investigators plan to reduce the amount of radiation treatment received to healthy tissue

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven tumors of the oral cavity, oropharynx, larynx, or hypopharynx .
* Treated with surgical resection with one (or both) side(s) of the neck pathologically N0.
* Indication for radiation therapy at the primary site or neck consisting of any of the below characteristics:

  * Close margin (<= 0.5 cm)
  * Positive margin
  * Perineural invasion
  * Lymphovascular space invasion
  * Metastatic disease in more than one lymph node
  * Metastatic disease in more than one lymph node group
  * Extracapsular extension in any lymph node
  * Constellation of factors considered to be at risk based on the multi-disciplinary tumor board discussion.
* Age >= 18.
* Patients must sign study specific, Institutional Review Board (IRB)-approved consent form.

Exclusion Criteria:

* Previous head and neck cancer other than non melanoma skin cancer.
* Previous head and neck surgery.
* Female patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-04-11 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Thorstad, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chao KS, Low DA, Perez CA, Purdy JA. Intensity-modulated radiation therapy in head and neck cancers: The Mallinckrodt experience. Int J Cancer. 2000 Apr 20;90(2):92-103. doi: 10.1002/(sici)1097-0215(20000420)90:23.0.co;2-9. PMID 10814959
- [Background] Chao KS, Ozyigit G, Tran BN, Cengiz M, Dempsey JF, Low DA. Patterns of failure in patients receiving definitive and postoperative IMRT for head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2003 Feb 1;55(2):312-21. doi: 10.1016/s0360-3016(02)03940-8. PMID 12527043
- [Background] Chao KS, Majhail N, Huang CJ, Simpson JR, Perez CA, Haughey B, Spector G. Intensity-modulated radiation therapy reduces late salivary toxicity without compromising tumor control in patients with oropharyngeal carcinoma: a comparison with conventional techniques. Radiother Oncol. 2001 Dec;61(3):275-80. doi: 10.1016/s0167-8140(01)00449-2. PMID 11730997
- [Background] Chao KS, Deasy JO, Markman J, Haynie J, Perez CA, Purdy JA, Low DA. A prospective study of salivary function sparing in patients with head-and-neck cancers receiving intensity-modulated or three-dimensional radiation therapy: initial results. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):907-16. doi: 10.1016/s0360-3016(00)01441-3. PMID 11240231
- [Background] Ang KK, Trotti A, Brown BW, Garden AS, Foote RL, Morrison WH, Geara FB, Klotch DW, Goepfert H, Peters LJ. Randomized trial addressing risk features and time factors of surgery plus radiotherapy in advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):571-8. doi: 10.1016/s0360-3016(01)01690-x. PMID 11597795
- [Background] O'Sullivan B, Warde P, Grice B, Goh C, Payne D, Liu FF, Waldron J, Bayley A, Irish J, Gullane P, Cummings B. The benefits and pitfalls of ipsilateral radiotherapy in carcinoma of the tonsillar region. Int J Radiat Oncol Biol Phys. 2001 Oct 1;51(2):332-43. doi: 10.1016/s0360-3016(01)01613-3. PMID 11567806
- [Background] Jackson SM, Hay JH, Flores AD, Weir L, Wong FL, Schwindt C, Baerg B. Cancer of the tonsil: the results of ipsilateral radiation treatment. Radiother Oncol. 1999 May;51(2):123-8. doi: 10.1016/s0167-8140(99)00051-1. PMID 10435802
- [Background] Brazilian Head and Neck Cancer Study Group. End results of a prospective trial on elective lateral neck dissection vs type III modified radical neck dissection in the management of supraglottic and transglottic carcinomas. Head Neck. 1999 Dec;21(8):694-702. doi: 10.1002/(sici)1097-0347(199912)21:83.0.co;2-b. PMID 10562681
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Perez CA, Carmichael T, Devineni VR, Simpson JR, Frederickson J, Sessions D, Spector G, Fineberg B. Carcinoma of the tonsillar fossa: a nonrandomized comparison of irradiation alone or combined with surgery: long-term results. Head Neck. 1991 Jul-Aug;13(4):282-90. doi: 10.1002/hed.2880130404. PMID 1907952
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on 04/11/2007 and closed to accrual 04/07/2014.
Groups:
- Arm 1: Intensity Modulated Radiation Therapy (IMRT): -This study provides guidelines for volume to be contoured during IMRT based on tumor site and stage of tumor site. The clinical tumor volume (CTV)1 will be treated to 66 Cy in 33 fractions or 60 Gy in 30 fractions. The CTV2 will be treated to 54 Gy in 33 fractions or 52 Gy in 30 fractions. The CTV3 will be modified based on tumor site and stage of tumor site in order to reduce volume.
Period: Overall Study
Arm/Group | Arm 1: Intensity Modulated Radiation Therapy (IMRT)
Started | 73
Completed | 72
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Intensity Modulated Radiation Therapy (IMRT)
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 56 [31 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 59
Region of Enrollment [Number; unit: participants]
  United States | 73
Primary tumor type [Number; unit: participants]
  Oropharynx | 37
  Larynx | 17
  Oral cavity | 14
  Hypopharynx | 4
  Unknown | 1
Tobacco abuse [Number; unit: participants]
  Yes | 47
  No | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Recurrence in the Unirradiated Neck(s)
Description: * Recurrence in a PN0 neck that was not treated is the critical endpoint in this study.
  * Recurrence is defined as the return of cancer after treatment
  * Recurrence is determined by a CT, PET/CT, or MRI and it will be fused with the original treatment planning CT scan. This will allow correlation between the original dose distribution and contours with any recurrent disease.
Time Frame: 12 months of follow-up
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Arm 1: IMRT: CTV1 = 66 Gy in 33 fractions
  CTV2 = 60 Gy in 33 fractions
  CTV3 = 56 Gy in 33 fractions
  CTV3 Proto = 56 Gy in 33 fractions
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 72
participants | 0 [0 to 4.2]

2. Secondary Outcome: Kaplan Meier Estimate of Locoregional Recurrence Free Survival
Description: * Recurrence is defined as the return of cancer after treatment
  * Kaplan Meier Estimate of the percentage of participants whose cancer has not returned locoregionally in the specified time frame
Time Frame: 3 years
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 34
percentage of participants-Kaplan Meier | 88.6

3. Secondary Outcome: Quality of Life (QOL) as Measured by Overall Global QOL Scores
Description: -The Quality of Life (QOL) Evaluation (Swallowing and Dryness Questionnaire) will be used. 20 questions with answers of Strongly Agree to Strongly Disagree. Global score was scaled for a total score from 0 to 100 with 0 being the worst QOL and 100 the best QOL.
Time Frame: Median follow-up was 22 months
Population: 65 out of 73 patients had evaluable QOL data in Arm 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 65
units on a scale | 59.1410 (34.8294)

4. Secondary Outcome: Quality of Life (QOL) as Measured by Xerostomia QOL Data
Description: -The Quality of Life (QOL) Evaluation (Swallowing and Dryness Questionnaire) will be used. 20 questions with answers of Strongly Agree to Strongly Disagree. Xerostomia score was scaled for a total xerostomia score from 0 to 100 with 0 being the worst QOL and 100 the best QOL.
Time Frame: Median follow-up was 22 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 65
units on a scale | 39.5584 (26.0941)

5. Secondary Outcome: Compare Standard Treatment Volume (CTV and PTV) With Protocol Defined Treatment Volume in Terms of Organ Specific Dose Volume Histograms
Time Frame: Completion of follow-up (minimum of 5 years from completion of treatment)
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: Disease Specific Survival Rate
Time Frame: Completion of follow-up (minimum of 5 years from completion of treatment)
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Kaplan Meier Estimate of Overall Survival
Time Frame: 3 years
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 45
percentage of participants-Kaplan Meier | 75.8

8. Secondary Outcome: Patterns of Failure Associated With Implementation of Primary Objective
Description: For patients who demonstrate a local failure during follow-up, a computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imagine (MRI) scan is fused with the original treatment planning CT scan using the computational environment for radiation research (CERR) developed at Washington University Medical Center. The methodology to transfer the digital imaging study via network to the radiation therapy research servers is mature. The original dose distribution and contours are correlated with the recurrent disease noted on the follow up imaging study. The recurrence is then classified as infield, marginal to the treatment field, or out of the treatment field depending on the dose received by the recurrent disease. Failures that occur in the treatment field are due to aspects of tumor biology rather than errors in the volume irradiated. As has been the case in our historical controls, the investigators expect most failures to be in the treatment field.
Time Frame: Completion of follow-up (minimum of 5 years from completion of treatment)
Reporting Status: Not Posted, anticipated posting 2026-04

9. Post Hoc Outcome: Kaplan Meier Estimate of Regional Recurrence Free Survival
Description: -Recurrence is defined as the return of cancer after treatment
Time Frame: 3 years
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 31
percentage of participants-Kaplan Meier | 94.8

10. Post Hoc Outcome: Kaplan Meier Estimate of Progression-free Survival
Description: -Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST 1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 3 years
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Arm 1: IMRT
Number analyzed (Participants) | 49
percentage of participants-Kaplan Meier | 68.9

ADVERSE EVENTS:
Arm/Group | Arm 1: Intensity Modulated Radiation Therapy (IMRT)
Serious Adverse Events (participants affected / at risk) | 7/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Intensity Modulated Radiation Therapy (IMRT) (N=72)
Death NOS (General disorders) | 1
Edema: head and neck (General disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Dyspnea (Gastrointestinal disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 2
Psychosis (Psychiatric disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Platelets (Investigations) | 1
Fever (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infection - catheter (Infections and infestations) | 1
Mucositis - oral cavity (Gastrointestinal disorders) | 2
Rash (erythema) (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Oral cavity pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Generalized weakness (General disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Intensity Modulated Radiation Therapy (IMRT) (N=72)
ALT, SGPT (Investigations) | 1
ALT, SGPT (late radiation morbidity) (Investigations) | 4
ANC/Neutrophils (late radiation morbidity) (Investigations) | 1
AST, SGOT (Investigations) | 1
AST, SGOT (late radiation morbidity) (Investigations) | 3
Abdomen pain (late radiation morbidity) (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Albumin (late radiation morbidity) (Metabolism and nutrition disorders) | 6
Albumin, serum-low (Metabolism and nutrition disorders) | 3
Alkaline phosphatase (Investigations) | 2
Allergic rhinitis (Immune system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Anorexia (late radiation morbidity) (Metabolism and nutrition disorders) | 2
Apnea (late radiation morbidity) (Nervous system disorders) | 1
Arm pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration pneumonia secondary to squamous cell carcinoma (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 4
Bilirubin (late radiation morbidity) (Investigations) | 1
Calcium, serum-high (Metabolism and nutrition disorders) | 1
Calcium, serum-low (Metabolism and nutrition disorders) | 8
Calcium, serum-low (late radiation morbidity) (Metabolism and nutrition disorders) | 5
Calcium, serum-low (late radiation morbidity) (Metabolism and nutrition disorders) | 2
Cardiac arrest (late radiation morbidity) (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Chest/thorax NOS pain (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 2
Clavicle pain (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 1
Cognitive disturbance (late radiation morbidity) (Nervous system disorders) | 1
Confusion (late radiation morbidity) (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Constipation (late radiation morbidity) (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cough (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 8
Creatinine (Investigations) | 4
Creatinine (late radiation morbidity) (Investigations) | 1
Death NOS (late radiation morbidity) (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Diarrhea (late radiation morbidity) (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 1
Dizziness (late radiation morbidity) (Nervous system disorders) | 2
Dry mouth (late radiation morbidity) (Gastrointestinal disorders) | 28
Dry mouth/salivary gland (Gastrointestinal disorders) | 23
Dysphagia (Gastrointestinal disorders) | 33
Dysphagia (late radiation morbidity) (Gastrointestinal disorders) | 26
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 3
Ear hemorrhage/bleeding (Ear and labyrinth disorders) | 1
Ear pain (late radiation morbidity) (Ear and labyrinth disorders) | 1
Edema: head and neck (General disorders) | 21
Edema: head and neck (late radiation morbidity) (General disorders) | 18
Edema: larynx (Respiratory, thoracic and mediastinal disorders) | 3
Edema: limb (late radiation morbidity) (General disorders) | 1
Edema: oropharynx (General disorders) | 2
Erythema (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 3
Esophagitis (Gastrointestinal disorders) | 2
Face pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 1
Failure to thrive (General disorders) | 1
Fatigue (General disorders) | 18
Fatigue (late radiation morbidity) (General disorders) | 12
Fever (General disorders) | 3
Fever (late radiation morbidity) (General disorders) | 1
Fistula (late radiation morbidity) (Gastrointestinal disorders) | 1
Generalized pain (General disorders) | 9
Glucose, serum-high (Metabolism and nutrition disorders) | 3
Glucose, serum-high (late radiation morbidity) (Metabolism and nutrition disorders) | 3
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 4
Hair loss/alopecia (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 1
Headache (late radiation morbidity) (Nervous system disorders) | 4
Hearing (Ear and labyrinth disorders) | 3
Hearing (late radiation morbidity) (Ear and labyrinth disorders) | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 24
Hemoglobin (late radiation morbidity) (Blood and lymphatic system disorders) | 14
Hemorrhage pulmonary/upper respiratory (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage, oral cavity (late radiation morbidity) (Gastrointestinal disorders) | 1
Hemorrhoids (late radiation morbidity) (Gastrointestinal disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Hypertension (late radiation morbidity) (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
INR (Investigations) | 1
INR (late radiation morbidity) (Investigations) | 6
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 2
Induration/fibrosis (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 2
Infection with normal ANC or grade 1 or 2 neutrophils (Infections and infestations) | 2
Insomnia (late radiation morbidity) (Psychiatric disorders) | 1
Jaw pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 3
Joint function (stiff) (Musculoskeletal and connective tissue disorders) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Leukocytes (late radiation morbidity) (Investigations) | 4
Leukocytes (total WBC) (Investigations) | 17
Libido (late radiation morbidity) (Reproductive system and breast disorders) | 1
Limb pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 1
Lymphopenia (Investigations) | 27
Lymphopenia (late radiation morbidity) (Investigations) | 17
Magnesium, serum-low (Metabolism and nutrition disorders) | 1
Metastatic disease (late radiation morbidity) (General disorders) | 4
Mood alteration: anxiety (Psychiatric disorders) | 3
Mood alteration: anxiety (late radiation morbidity) (Psychiatric disorders) | 2
Mood alteration: depression (Psychiatric disorders) | 7
Mood alteration: depression (late radiation morbidity) (Psychiatric disorders) | 6
Mouth (thrush) infection (late radiation morbidity) (Infections and infestations) | 1
Mucositis (late radiation morbidity) (Gastrointestinal disorders) | 1
Mucositis - oral cavity (Gastrointestinal disorders) | 41
Mucositis - oropharynx (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional) (Gastrointestinal disorders) | 12
Mucositis/stomatitis - oral cavity (late radiation morbidity) (Gastrointestinal disorders) | 8
Muscle weakness (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 23
Nausea (late radiation morbidity) (Gastrointestinal disorders) | 7
Neck fistula (late radiation morbidity) (Gastrointestinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 11
Neck pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 14
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 5
Neuropathy: sensory (late radiation morbidity) (Nervous system disorders) | 4
Neutrophils/Granulocytes (Investigations) | 9
Obstruction (late radiation morbidity) (Gastrointestinal disorders) | 1
Oral cavity fibrosis (tongue) (late radiation morbidity) (Gastrointestinal disorders) | 2
Oral cavity pain (Gastrointestinal disorders) | 11
Oral cavity pain (late radiation morbidity) (Gastrointestinal disorders) | 4
Oropharynx pain (Respiratory, thoracic and mediastinal disorders) | 5
Osteoradionecrosis (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 1
PTT (late radiation morbidity) (Investigations) | 1
Pericarditis (Cardiac disorders) | 1
Pharynx pain (Respiratory, thoracic and mediastinal disorders) | 3
Platelets (Investigations) | 7
Platelets (late radiation morbidity) (Investigations) | 2
Pneumonia (Infections and infestations) | 3
Pneumonia (late radiation morbidity) (Infections and infestations) | 1
Potassium (late radiation morbidity) (Metabolism and nutrition disorders) | 5
Potassium, serum-high (Metabolism and nutrition disorders) | 1
Potassium, serum-low (late radiation morbidity) (Metabolism and nutrition disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Radiation changes - pharynx/esophagus (Injury, poisoning and procedural complications) | 2
Rash - dermatitis (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 8
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation (Injury, poisoning and procedural complications) | 23
Rigors/chills (late radiation morbidity) (Investigations) | 1
Salivary gland changes, saliva (late radiation morbidity) (Gastrointestinal disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 15
Salivary glands (late radiation morbidity) (Gastrointestinal disorders) | 3
Shoulder pain (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 2
Skin (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 3
Skin changes (Skin and subcutaneous tissue disorders) | 2
Skin tightness (late radiation morbidity) (Skin and subcutaneous tissue disorders) | 1
Sodium, serum-high (late radiation morbidity) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (Metabolism and nutrition disorders) | 2
Sodium, serum-low (late radiation morbidity) (Metabolism and nutrition disorders) | 4
Somnolence/depressed level of consciousness (Nervous system disorders) | 2
Speech impairment (Nervous system disorders) | 5
Speech impairment (late radiation morbidity) (Nervous system disorders) | 1
Syncope (late radiation morbidity) (Nervous system disorders) | 2
Taste alteration (Gastrointestinal disorders) | 23
Teeth discoloration (late radiation morbidity) (Gastrointestinal disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Throat/larynx pain (Respiratory, thoracic and mediastinal disorders) | 7
Throat/pharynx/larynx pain (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 7
Thrombosis/thrombus/embolism (late radiation morbidity) (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 4
Tongue pain (late radiation morbidity) (Gastrointestinal disorders) | 1
Tracheitis (late radiation morbidity) (Infections and infestations) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Trismus (late radiation morbidity) (Musculoskeletal and connective tissue disorders) | 3
Upper respiratory infection (late radiation morbidity) (Infections and infestations) | 1
Vision-blurred vision (late radiation morbidity) (Eye disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 17
Voice changes/dysarthria (late radiation morbidity) (Respiratory, thoracic and mediastinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 16
Vomiting (late radiation morbidity) (Gastrointestinal disorders) | 5
Watery eye (Eye disorders) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 24
Weight loss (late radiation morbidity) (General disorders) | 8
Wound complication, non infectious (late radiation morbidity) (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes